CLINICAL TRIAL: NCT06364228
Title: Intranasal Oxytocin Intervention for Caregivers to Persons With Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0133-24-FB
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-07

CONDITIONS: Stress
Keywords: Oxytocin; Stress level; Caregivers; Dementia; fMRI; Neuroimaging; Quality of Life
MeSH Terms: conditions — Dementia | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intranasal Spray Placebo (Placebo Comparator): Nasal spray of placebo liquid solution is administered as 2 puffs of daily dose (every morning) for 3 weeks. Functional magnetic resonance imaging (fMRI) scan will be done pre- and post-administration.
  Interventions: Drug: Placebo; Procedure: Functional MRI
- Oxytocin Intranasal Spray 12 International Units (Active Comparator): Nasal spray of Oxytocin 12 International Units (12IU) liquid solution as 2 puffs of daily dose (every morning) for 3 weeks. Functional magnetic resonance imaging (fMRI) scan pre- and post-administration.
  Interventions: Drug: Oxytocin Intranasal Spray 12 International Unit (12IU); Procedure: Functional MRI
- Oxytocin Intranasal Spray 24 International Units (Active Comparator): Nasal spray of Oxytocin 24 International Units (24IU) liquid solution as 2 puffs of daily dose (every morning) for 3 weeks. Functional magnetic resonance imaging (fMRI) scan pre- and post-administration.
  Interventions: Drug: Oxytocin Intranasal Spray 24 International Unit (24IU); Procedure: Functional MRI

INTERVENTIONS:
Drug: Placebo — Placebo intranasal spray liquid with no oxytocin will be delivered in 2 puffs to each nostril daily for 21 days. The first single dose will be administered at the clinic (Visit 1).
  Arms: Intranasal Spray Placebo
Drug: Oxytocin Intranasal Spray 12 International Unit (12IU) — Participants weighing less than 40 kg (88 pounds) will receive 12 IU of oxytocin delivered as 1 puff (6 IU) to each nostril daily for 21 days. The first single dose will be administered at the clinic (Visit 1).
  Other Names: Oxytocin 12IU
  Arms: Oxytocin Intranasal Spray 12 International Units
Drug: Oxytocin Intranasal Spray 24 International Unit (24IU) — Participants weighing more than 40 kg (880 pounds) will receive 24 IU of oxytocin delivered as 2 puffs (12 IU) to each nostril daily for 21 days. The first single dose will be administered at the clinic (Visit 1).
  Other Names: Oxytocin 24IU
  Arms: Oxytocin Intranasal Spray 24 International Units
Procedure: Functional MRI — Functional MRI (fMRI) scan with affective Stroop and Empathy and Theory of Mind task (EmpaTom task will administered pre- and post-administration of oxytocin.
  Other Names: fMRI

SUMMARY:
More than 15 million family caregivers provide support for individuals with Alzheimer's disease (AD) or related dementias. This number is expected to grow with the increasing population of persons with dementia (PWD). Stress in caregivers to older adults with chronic diseases is already a significant public health issue because it is associated with multiple negative physical and mental health outcomes for the caregiver (e.g., depression, cardiovascular disease) and can negatively impact the health of the PWD as well. Importantly, stress levels are even higher in female than male caregivers and in caregivers to PWD than other chronic conditions that affect older adults.

There are numerous interventions to improve well-being in caregivers to PWD, but only two have been shown to moderately improve caregiver depression and quality of life in the PWD. However, both of the interventions are time and energy intensive. One promising candidate to reduce stress and improve quality of life is the endogenous neuropeptide oxytocin (OXT). Intranasal OXT interventions have been shown to successfully reduce stress and increase quality of life in other populations, including patients with borderline personality disorder, Post-traumatic Stress Disorder (PTSD), Anxiety Disorder, and Depressive Disorder. This study will assess the efficacy and safety of intranasal oxytocin (OXT) to improve the quality of life and reduce chronic stress levels in the caregivers to PWD. Participants will be randomly enrolled to one of three groups: 12 IU intranasal oxytocin, 24 IU intranasal oxytocin or placebo. The study drug will be administered daily for 21 days.

DETAILED DESCRIPTION:
More than 15 million family caregivers provide support for individuals with Alzheimer's disease (AD) or related dementias. This number is expected to grow with the increasing population of persons with dementia (PWD). Stress in caregivers to older adults with chronic diseases is already a significant public health issue because it is associated with multiple negative physical and mental health outcomes for the caregiver (e.g., depression, cardiovascular disease) and can negatively impact the health of the PWD as well. Importantly, stress levels are even higher in female than male caregivers and in caregivers to a PWD than other chronic conditions that affect older adults. One promising candidate to reduce stress and improve quality of life is the endogenous neuropeptide oxytocin (OXT). Intranasal OXT interventions have been shown to successfully reduce stress and increase quality of life in other populations, including patients with borderline personality disorder, Post-traumatic Stress Disorder (PTSD), Anxiety Disorder, and Depressive Disorder. However, currently there is no comprehensive study examining its role in the caregivers to chronic medical/psychiatric illnesses including dementia for potential beneficial impact as well as reducing chronic stress levels.

Eligible females who are family caregivers to a PWD for a least five hours a week for six consecutive months will be randomly enrolled to one of three groups: 12 IU intranasal oxytocin, 24 IU intranasal oxytocin or placebo. The study drug will be administered daily for 21 days. Surveys and questionnaires that evaluate mental and emotional health and functional magnetic resonance imaging (fMRI) will be administered before and after the study treatment to see if oxytocin will help improve quality of life better and lower stress levels in caregivers to people who have dementia. Additionally, the study will find out if the brain responds to oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* Females 50 years of age or older
* Currently an unpaid family caregiver to an older adult (50 years and older) with dementia for at least five hours a week for at least six months
* Normal or corrected to normal vision and hearing
* Mobility to travel to University of Nebraska Medical Center (UNMC) for study procedures including brain imaging
* Right-handed
* Capacity to read and write English

Exclusion Criteria:

* Major medical illness that contraindicates oxytocin (OXT) administration (e.g., severe liver disease, seizure disorder, metabolic disorder)
* History of allergic reaction to oxytocin (OXT) and its nasal spray product
* History of central nervous system (CNS) disease, including history of seizure, epilepsy, CNS tumor, CNS hemorrhage, or serious CNS infection including meningitis or encephalitis
* Currently pregnant or planning to become pregnant during the course of the study
* Metal in the body (i.e., hearing aid, cardiac pacemaker, bone plates, braces, non-removable piercing/implants, etc.), claustrophobia, or any other condition that would preclude magnetic resonance imaging (MRI) scanning
* Mini-mental status exam score of 25 or lower which suggests possible cognitive issues
* History of or current neurological disease (e.g., stroke, traumatic brain injury, brain tumor, dementia)
* History of or current severe psychiatric disease (e.g., schizophrenia, bipolar disorder, autism, severe post-traumatic stress disorder)
* History of, or current drug or alcohol abuse
* Currently breastfeeding
* Current coronavirus disease-19 (COVID-19) illness
* Left-handed due to brain structural difference between right and left-handed individuals
* Currently taking antipsychotic medications, selective serotonin reuptake inhibitors (SSRIs) or corticosteroid creams/pills

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Chronic Stress Level in the Past Thirty Days | Baseline (Visit 1) and Post-intervention (Visit 2)
  Participant's chronic ctress levels in the past thirty Days will be assessed by the Perceived Stress Scale (PSS) which asks ten questions about participant stress within the last 30 days. The questions are scored from 0 ("never") to 4 ("very often) with specific items needing to be reverse scored. Higher scores indicate higher levels of perceived stress (a worse outcome). The instrument takes about 5 minutes to complete.

SECONDARY OUTCOMES:
Participant Quality of Life | Baseline (Visit 1) and Post-intervention (Visit 2)
  Participant quality of life will be assessed by the Health Organization Quality of Life- Short version (WHO-QOL-BREF) survey which measures general perceptions about quality of life in four aspects: physical health, psychological health, social relationships, and environment. The aspects are scored from 1 ('very poor') to 5 ('very good'). Aspect scores are totaled with higher scores indicating a better outcome. The instrument takes about 15 minutes to complete.
Blood Oxygen Level Dependent (BOLD) responses in neural areas during the Affective Stroop task (AS) and Empathy and Theory of Mind(EmpaToM) task | Baseline (Visit 1) and Post-intervention (Visit 2) It will take about 60 minutes to complete at each time point.
  Neural level changes will be measured by Functional Magnetic Resonance Imaging (fMRI).

OTHER OUTCOMES:
Cognitive Orientation Screening | Visit 1 (Baseline visit). It will take about 10 minutes.
  Participants will complete a brief cognitive orientation screening tool, called the Mini-Mental Status Exam. This will be administered by the research assistant. If the participant scores below 26 on this measure, they will be excluded from the study, as it may indicate potential cognitive issues. The scale ranges from 0 to 30, with higher scores indicating better cognitive performance (better outcomes).
Geriatric Anxiety Scale (GAS-10) | Baseline (Visit 1) and Post-intervention (Visit 2) It will take about 5 minutes to complete at each time point.
  Geriatric Anxiety Scale (GAS-10) will assess 10 Items. The rating scale ranges from 0 to 30 points. Higher scores indicate more severe anxiety (worse outcomes).
Geriatric Depression Scale Short Form (GDS-SF) | Baseline (Visit 1) and Post-intervention (Visit 2) It will take about 7 minutes to complete at each time point.
  Geriatric Depression Scale Short Form (GDS-SF) is a rating scale from 0 to 15 points. Higher scores indicate more likelihood of depression symptoms and need for further assessment of depression (worse outcomes).
Alcohol Use Disorders Identification Test | Baseline (Visit 1) and Post-intervention (Visit 2)
  The Alcohol Use Disorders Identification Test (AUDIT Alcohol Screening Tool) assesses 10 items about alcohol consumption, drinking behaviors, and alcohol-related problems of the caregiver. Total scores range from 0 to 40. Higher scores indicate a greater likelihood of harmful alcohol consumption (worse outcomes). Caregivers will complete the instrument twice, each time taking about 10 minutes to finish.
Neuropsychiatric Inventory-Questionnaire | Baseline (Visit 1) and Post-intervention (Visit 2)
  The Neuropsychiatric Inventory-Questionnaire (NPI-Q) measures 12 domains. The caregiver selects present or absent for symptoms in each domain of the individual with dementia, then rates the severity of symptoms present in the past month. Each domain is scored from 0 to 3 and all domain scores are totaled. Higher scores indicating more severe symptoms (worse outcomes). This instrument also rates impact of the symptoms of individual with dementia on the caregiver (Distress) in each domain. The Distress of each domain is scored from 0 to 5 and all domain scores are totaled. Higher scores indicating more extreme levels of distress (worse outcomes). Caregivers will complete the instrument twice, each time taking about 5 minutes to finish.
Quick Dementia Rating Scale | Baseline (Visit 1) and Post-intervention (Visit 2)
  The Quick Dementia Rating Scale (QDRS) measures 10 different domains of daily functioning, mood, and behavior. Caregivers rate the severity of dementia symptoms in each domain about the individual for whom they are providing care. Total scores range from 0 to 30, with higher scores indicating more impairment (worse outcomes). Caregivers will complete the instrument twice, each time taking about 5 minutes to finish.
The Interpersonal Reactivity Index | Baseline (Visit 1) and Post-intervention (Visit 2)
  The Interpersonal Reactivity Index (IRI) is a multidimensional measure of empathy of the caregiver. This instrument has four subscales: Perspective Taking, Empathic Concern, Personal Distress, and Fantasy. Each subscale has 7 items scored from 0 to 4 with specific items needing to be reverse scored. Higher scores indicate greater empathy (better outcomes). Caregivers will complete the instrument twice, each time taking about 10 minutes to finish.

CONTACTS AND LOCATIONS:
Overall Officials: Soonjo Hwang, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Psychiatry, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimers Association. 2015 Alzheimers Disease Facts and Figures. (2015).
- [Background] Pinquart M, Sorensen S. Differences between caregivers and noncaregivers in psychological health and physical health: a meta-analysis. Psychol Aging. 2003 Jun;18(2):250-67. doi: 10.1037/0882-7974.18.2.250. PMID 12825775
- [Background] Peavy G, Mayo AM, Avalos C, Rodriguez A, Shifflett B, Edland SD. Perceived Stress in Older Dementia Caregivers: Mediation by Loneliness and Depression. Am J Alzheimers Dis Other Demen. 2022 Jan-Dec;37:15333175211064756. doi: 10.1177/15333175211064756. PMID 34986661
- [Background] Sheehan OC, Haley WE, Howard VJ, Huang J, Rhodes JD, Roth DL. Stress, Burden, and Well-Being in Dementia and Nondementia Caregivers: Insights From the Caregiving Transitions Study. Gerontologist. 2021 Jul 13;61(5):670-679. doi: 10.1093/geront/gnaa108. PMID 32816014
- [Background] Bouchard K, Greenman PS, Pipe A, Johnson SM, Tulloch H. Reducing Caregiver Distress and Cardiovascular Risk: A Focus on Caregiver-Patient Relationship Quality. Can J Cardiol. 2019 Oct;35(10):1409-1411. doi: 10.1016/j.cjca.2019.05.007. Epub 2019 Sep 9. PMID 31515084
- [Background] Losada-Baltar A, Vara-Garcia C, Pedroso-Chaparro MDS, Cabrera I, Jimenez-Gonzalo L, Fernandes-Pires J, Huertas-Domingo C, Barrera-Caballero S, Gallego-Alberto L, Romero-Moreno R, Marquez-Gonzalez M. Family caregivers of people with dementia in the context of the sociocultural stress and coping model: An examination of gender differences. J Women Aging. 2023 Jul-Aug;35(4):354-368. doi: 10.1080/08952841.2022.2052705. Epub 2022 Mar 26. PMID 35343403
- [Background] Riffin C, Van Ness PH, Wolff JL, Fried T. Multifactorial Examination of Caregiver Burden in a National Sample of Family and Unpaid Caregivers. J Am Geriatr Soc. 2019 Feb;67(2):277-283. doi: 10.1111/jgs.15664. Epub 2018 Nov 19. PMID 30452088
- [Background] Marques MJ, Tan EYL, Woods B, Jelley H, Kerpershoek L, Hopper L, Irving K, Bieber A, Stephan A, Skoldunger A, Sjolund BM, Selbaek G, Rosvik J, Zanetti O, Portolani DM, Maroco J, de Vugt M, Verhey F, Goncalves-Pereira M; Actifcare Consortium. Trajectories of relationship quality in dementia: a longitudinal study in eight European countries. Aging Ment Health. 2022 Nov;26(11):2307-2315. doi: 10.1080/13607863.2021.1969641. Epub 2021 Sep 6. PMID 34486887
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Care Services; Board on Health Sciences Policy; Committee on Care Interventions for Individuals with Dementia and Their Caregivers; Stroud C, Larson EB, editors. Meeting the Challenge of Caring for Persons Living with Dementia and Their Care Partners and Caregivers: A Way Forward. Washington (DC): National Academies Press (US); 2021 Feb 23. Available from http://www.ncbi.nlm.nih.gov/books/NBK567818/ PMID 33625814
- [Background] Butler M, et al. Care Interventions for People Living With Dementia and Their Caregivers. Comparative Effectiveness Review No. 231. (Prepared by the Minnesota Evidence-based Practice Center under Contract No. 290-2015-00008-I.) AHRQ Publication No. 20-EHC023. Rockville, MD: Agency for Healthcare Research and Quality; August 2020. Errata December 2020. DOI: https://doi.org/10.23970/AHRQEPCCER231.
- [Background] Cochran DM, Fallon D, Hill M, Frazier JA. The role of oxytocin in psychiatric disorders: a review of biological and therapeutic research findings. Harv Rev Psychiatry. 2013 Sep-Oct;21(5):219-47. doi: 10.1097/HRP.0b013e3182a75b7d. PMID 24651556
- [Background] Viero C, Shibuya I, Kitamura N, Verkhratsky A, Fujihara H, Katoh A, Ueta Y, Zingg HH, Chvatal A, Sykova E, Dayanithi G. REVIEW: Oxytocin: Crossing the bridge between basic science and pharmacotherapy. CNS Neurosci Ther. 2010 Oct;16(5):e138-56. doi: 10.1111/j.1755-5949.2010.00185.x. Epub 2010 Jul 7. PMID 20626426
- [Background] Simeon D, Bartz J, Hamilton H, Crystal S, Braun A, Ketay S, Hollander E. Oxytocin administration attenuates stress reactivity in borderline personality disorder: a pilot study. Psychoneuroendocrinology. 2011 Oct;36(9):1418-21. doi: 10.1016/j.psyneuen.2011.03.013. Epub 2011 May 4. PMID 21546164
- [Background] Olff M, Frijling JL, Kubzansky LD, Bradley B, Ellenbogen MA, Cardoso C, Bartz JA, Yee JR, van Zuiden M. The role of oxytocin in social bonding, stress regulation and mental health: an update on the moderating effects of context and interindividual differences. Psychoneuroendocrinology. 2013 Sep;38(9):1883-94. doi: 10.1016/j.psyneuen.2013.06.019. Epub 2013 Jul 12. PMID 23856187
- [Background] De Cagna F, Fusar-Poli L, Damiani S, Rocchetti M, Giovanna G, Mori A, Politi P, Brondino N. The Role of Intranasal Oxytocin in Anxiety and Depressive Disorders: A Systematic Review of Randomized Controlled Trials. Clin Psychopharmacol Neurosci. 2019 Feb 28;17(1):1-11. doi: 10.9758/cpn.2019.17.1.1. PMID 30690935
- [Background] Arueti M, Perach-Barzilay N, Tsoory MM, Berger B, Getter N, Shamay-Tsoory SG. When two become one: the role of oxytocin in interpersonal coordination and cooperation. J Cogn Neurosci. 2013 Sep;25(9):1418-27. doi: 10.1162/jocn_a_00400. Epub 2013 Apr 11. PMID 23574582
- [Background] Levy J, Goldstein A, Zagoory-Sharon O, Weisman O, Schneiderman I, Eidelman-Rothman M, Feldman R. Oxytocin selectively modulates brain response to stimuli probing social synchrony. Neuroimage. 2016 Jan 1;124(Pt A):923-930. doi: 10.1016/j.neuroimage.2015.09.066. Epub 2015 Oct 9. PMID 26455794
- [Background] Grace SA, Rossell SL, Heinrichs M, Kordsachia C, Labuschagne I. Oxytocin and brain activity in humans: A systematic review and coordinate-based meta-analysis of functional MRI studies. Psychoneuroendocrinology. 2018 Oct;96:6-24. doi: 10.1016/j.psyneuen.2018.05.031. Epub 2018 May 24. PMID 29879563
- [Background] Kendrick KM, Guastella AJ, Becker B. Overview of Human Oxytocin Research. Curr Top Behav Neurosci. 2018;35:321-348. doi: 10.1007/7854_2017_19. PMID 28864976
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Mueller AE, Segal DL, Gavett B, Marty MA, Yochim B, June A, Coolidge FL. Geriatric Anxiety Scale: item response theory analysis, differential item functioning, and creation of a ten-item short form (GAS-10). Int Psychogeriatr. 2015 Jul;27(7):1099-111. doi: 10.1017/S1041610214000210. Epub 2014 Feb 27. PMID 24576589
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Weintraub S, Salmon D, Mercaldo N, Ferris S, Graff-Radford NR, Chui H, Cummings J, DeCarli C, Foster NL, Galasko D, Peskind E, Dietrich W, Beekly DL, Kukull WA, Morris JC. The Alzheimer's Disease Centers' Uniform Data Set (UDS): the neuropsychologic test battery. Alzheimer Dis Assoc Disord. 2009 Apr-Jun;23(2):91-101. doi: 10.1097/WAD.0b013e318191c7dd. PMID 19474567
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Blair KS, Smith BW, Mitchell DG, Morton J, Vythilingam M, Pessoa L, Fridberg D, Zametkin A, Sturman D, Nelson EE, Drevets WC, Pine DS, Martin A, Blair RJ. Modulation of emotion by cognition and cognition by emotion. Neuroimage. 2007 Mar;35(1):430-40. doi: 10.1016/j.neuroimage.2006.11.048. Epub 2007 Jan 18. PMID 17239620
- [Background] Blair KS, Geraci M, Smith BW, Hollon N, DeVido J, Otero M, Blair JR, Pine DS. Reduced dorsal anterior cingulate cortical activity during emotional regulation and top-down attentional control in generalized social phobia, generalized anxiety disorder, and comorbid generalized social phobia/generalized anxiety disorder. Biol Psychiatry. 2012 Sep 15;72(6):476-82. doi: 10.1016/j.biopsych.2012.04.013. Epub 2012 May 15. PMID 22592057
- [Background] Lang PJ BM, Cuthbert BN. International affective picture system (IAPS): Affetive ratings of pictures and instruction manual. Gainesville, FL: University of Florida; 2005.
- [Background] Hwang S, Nolan ZT, White SF, Williams WC, Sinclair S, Blair RJ. Dual neurocircuitry dysfunctions in disruptive behavior disorders: emotional responding and response inhibition. Psychol Med. 2016 May;46(7):1485-96. doi: 10.1017/S0033291716000118. Epub 2016 Feb 15. PMID 26875722
- [Background] Hwang S, White SF, Nolan ZT, Craig Williams W, Sinclair S, Blair RJ. Executive attention control and emotional responding in attention-deficit/hyperactivity disorder--A functional MRI study. Neuroimage Clin. 2015 Oct 9;9:545-54. doi: 10.1016/j.nicl.2015.10.005. eCollection 2015. PMID 26640766
- [Background] Marsh AA, Finger EC, Mitchell DG, Reid ME, Sims C, Kosson DS, Towbin KE, Leibenluft E, Pine DS, Blair RJ. Reduced amygdala response to fearful expressions in children and adolescents with callous-unemotional traits and disruptive behavior disorders. Am J Psychiatry. 2008 Jun;165(6):712-20. doi: 10.1176/appi.ajp.2007.07071145. Epub 2008 Feb 15. PMID 18281412
- [Background] White SF, Marsh AA, Fowler KA, Schechter JC, Adalio C, Pope K, Sinclair S, Pine DS, Blair RJ. Reduced amygdala response in youths with disruptive behavior disorders and psychopathic traits: decreased emotional response versus increased top-down attention to nonemotional features. Am J Psychiatry. 2012 Jul;169(7):750-8. doi: 10.1176/appi.ajp.2012.11081270. PMID 22456823
- [Background] Kanske P, Bockler A, Trautwein FM, Singer T. Dissecting the social brain: Introducing the EmpaToM to reveal distinct neural networks and brain-behavior relations for empathy and Theory of Mind. Neuroimage. 2015 Nov 15;122:6-19. doi: 10.1016/j.neuroimage.2015.07.082. Epub 2015 Aug 5. PMID 26254589
- [Background] Galvin JE. THE QUICK DEMENTIA RATING SYSTEM (QDRS): A RAPID DEMENTIA STAGING TOOL. Alzheimers Dement (Amst). 2015 Jun 1;1(2):249-259. doi: 10.1016/j.dadm.2015.03.003. PMID 26140284
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Posner, K., Brent, D., Lucas, C., Gould, M., Stanley, B., Brown, G., Fisher, P., Zelazny, J., Burke, A., Oquendo, M., Mann, J. (2008). Columbia Suicide Severity Rating Scale (CSSRS) Since Last Visit. The Research Foundation for Mental Hygiene, Inc.